CLINICAL TRIAL: NCT05991037
Title: Consequence of Plasma Concentrations of Psychoactive Drugs Located Beyond Therapeutic Ranges on Severity of Falls in Patients Over 75 Years Old
Brief Title: Relation Between Psychoactive Drugs Overdosage and Severity of Falls in Elderly People
Acronym: MEDIFALL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-0177
Record Dates: First submitted 2022-08-23; First posted 2023-08-14 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Fall
Keywords: fall; psychoactive drugs; old patients; prescription; plasmatic concentrations
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: The severity of the fall will be assessed in the 400 patients included. The groups will be defined a posteriori, according to the results obtained for the psychoactive drug dosages.
  Approximately 80 patients expected in the "overdosed" group matched to the same number of subjects on gender, age and cognition from the 320 subjects in the "non-overdosed" group to meet the primary objective at risk α = 5% and a power = 80%.
Masking Description: The groups will be constituted after the inclusions according to the results of the psychoactive drug blood concentration measures, so that Participants, Care Provider and Investigators will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "overdosed" group (Experimental): The experimental group will be made up of falling patients recruited for whom at least one psychoactive drug has been measured in a concentration higher than the usual therapeutic ranges.
  Interventions: Biological: Blood sampling for psychoactive drugs dosage
- "non-overdosed" group (Other): The control group will be made up of falling patients recruited for whom none of the psychoactive drugs have been measured in supra-therapeutic concentrations (therefore concentrations measured therapeutic or infra-therapeutic)
  Interventions: Biological: Blood sampling for psychoactive drugs dosage

INTERVENTIONS:
Biological: Blood sampling for psychoactive drugs dosage — 4 blood samples for psychoactive drugs identification and dosage will be taken on arrival at the emergency room during fall management

SUMMARY:
There are many epidemiological data on the relationship between the number or nature of psychoactive medications used and the risk of falling in elderly, but very little on the relationship between the amount of psychoactive medication actually present in the blood and the severity of the fall. However, the inevitable drug-drug interactions related to polypharmacy and the pharmacokinetic modifications related to old age may lead plasma overdose situations which can potentiate the risk of falls but also aggravate these consequences. The investigators therefore propose a study with the objective of verifying whether the proportion of falls with serious traumatic consequences is more frequent in patients over 75 years old, presenting plasma overdoses of psychoactive drugs (plasma concentrations higher than the usual therapeutic concentrations) in regard to those between therapeutic ranges.

The aim of this work is to verify if the falls present more severe characters when the psychoactive drug concentrations are beyond the usual therapeutic ranges.

DETAILED DESCRIPTION:
Patients over the age of 75 with at least one psychoactive drugs in their usual treatment will be included in the study in order to assess the severity of their fall and to measure the concentrations of all psychoactive drugs identified in their blood samples.

This study must include 400 patients over the age of 75 hospitalized for a fall in geriatrics or another department after going to the emergency room.

Patients will be included in the study as soon as they go to the emergency room during which the blood samples will be taken and several data collected. The final inclusions and the consultations to collect the clinical and biological data essential to the achievement of the main and secondary objectives will then be carried out by a geriatrician in the patient's hospitalization department.

Qualitative research and plasma assays of psychoactive drugs will be carried out by liquid phase chromatography coupled with a tandem mass spectrometer.

The expected duration of the study will be 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient (male, female) aged 75 and over admitted to the emergency room for a fall and for whom hospitalization (in geriatrics or not) after going to the emergency room is planned
* Patient consuming at least one psychoactive drug from the list provided in the protocol
* Patient able to move before hospitalization with or without technical assistance
* Patient who signed the consent
* Patient subject to the social security system

Exclusion Criteria:

* Patient not requiring hospitalization after going to the emergency room
* Patient having fallen for more than 12 hours before inclusion in the study (time of sampling) [risk of excessive elimination of certain drugs with short half-lives]
* Parkinsonian patient or patient who has fallen following a convulsive attack
* Patient with a life-threatening prognosis in the very short term (state of shock, palliative care planned from the emergency room)
* Patient in wheelchair or bedridden
* Adult under legal protection, guardianship, curators
* Patient not understanding the French language

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of the percentages of falls with serious traumatic consequences in each of the two "overdosed" and "non-overdosed" groups. | 3 years
  To evaluate if serious traumatic consequences are more important in the group of elderly patients with plasma overdoses of psychoactive drugs than in the "non-overdosed" group.

SECONDARY OUTCOMES:
Relationship between the category of severity of the fall (according to the criteria of Schwenk et al, 2012) and the interactions highlighted in the prescription | 3 years
  To evaluate influence of prescribed medication on the nature of the fall.
  * Prescription prior to the fall will be evaluated taking into account the drug-drug interactions. This analysis will be done taking into account the number of interactions, the effect of interactions (increase, decrease or suppression of the effect), the level of recommendations (contraindication, not recommended, precaution for use, to be taken into account).
  * Severity of the fall will be evaluated according to the criteria of Schwenk et al, 2012 (serious, moderate, minor or no injuries).
Relationship between the blood concentrations of psychoactive drugs and the occurrence of confusional syndrome assessed by the Confusion Assessment Method and/or neurocognitive disorders assessed by the Mini Mental State Evaluation. | 3 years
  To evaluate influence of psychoactive drug overdosage on confusional and/or cognitive state
  * Blood concentrations of psychoactive drugs were measured by chromatographic methods with different unit of measure (mg/l; µg/l; mmol/l).
  * Confusion Assessment Method (CAM) with 3 mandatory criteria and 2 facultative criteria.
  * Mini Mental State Evaluation (MMSE) with total score between 0 and 30 (0 corresponding to severe impairment and 30 to no damage.
Relationship between drug blood concentrations and severity of the fall, various states and functions studied during the geriatric consultation (dependence, mood, nutritional state, renal and liver function, presence of drug-drug interactions). | 3 years
  To evaluate the influence of psychoactive drug blood concentrations on :
  * severity of the fall (same criteria as in Outcome 2)
  * dependence, evaluated with 2 scales: Instrumental Activities of Daily Living (IADL) scale ranging 0 (indicating complete dependence) to 8 (indicating complete autonomy) and Activities of Daily Living (ADL) scale ranging 0 (indicating complete dysautonomia) to 6 (indicating complete autonomy) ,
  * mood, evaluated with Geriatric Depression Scale (GDS) ranging 0 (as normal mood) to 15 (as high likelihood of depression)
  * nutritional status, evaluated with Body Mass Index (kg/m2) and albuminemia (g/L)
  * renal function evaluated with Chronic Kidney Disease EPIdemiology (CKD Epi) or Modification of Diet in Renal Disease (MDRD) (ml/min/1.73m2)
  * liver function, evaluated with liver enzymes measurement (alanine aminotransferase ALAT, aspartate transaminase ASAT IU/L),
  * presence of drug-drug interactions (same criteria as in Outcome 2)
Comparison between psychoactive drugs identified in the blood and expected prescriptions (entry prescription) | 3 years
  To evaluate the level of adequacy between the prescription (expected prescriptions, verification of misuse, compliance, etc.) and the psychoactive drugs (nature and quantity evaluated as in outcome 3) found in the blood by chromatographic method.
Evaluation of the severity of the fall (according to the criteria of Schwenk et al, 2012) with regard to a recent modification or not of the prescription (descriptive presentation of modification of dosage, addition ore deletion) | 3 years
  To evaluate the influence of recent change in the prescription (taking into account any recent adjustments to it: modification of dosage, addition of prescription or deletion of prescription) on the severity of the fall (criteria of Schwenk et al, 2012: serious, moderate, minor or no injuries).

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Lelong-Boulouard, PhD, Study Director — Caen Normandie Universitary Hospital Center
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No
All study data is the exclusive property of the Promoter. Any publication relating to these can only be made after validation by the Promoter and the lead methodologist.

REFERENCES:
- [Background] Bloch F, Thibaud M, Dugue B, Breque C, Rigaud AS, Kemoun G. Psychotropic drugs and falls in the elderly people: updated literature review and meta-analysis. J Aging Health. 2011 Mar;23(2):329-46. doi: 10.1177/0898264310381277. Epub 2010 Oct 14. PMID 20947876
- [Background] Han JH, Chen A, Vasilevskis EE, Schnelle JF, Ely EW, Chandrasekhar R, Morrison RD, Ryan TP, Daniels JS, Sutherland JJ, Simmons SF. Supratherapeutic Psychotropic Drug Levels in the Emergency Department and Their Association with Delirium Duration: A Preliminary Study. J Am Geriatr Soc. 2019 Nov;67(11):2387-2392. doi: 10.1111/jgs.16156. Epub 2019 Sep 10. PMID 31503339
- [Background] Schwenk M, Lauenroth A, Stock C, Moreno RR, Oster P, McHugh G, Todd C, Hauer K. Definitions and methods of measuring and reporting on injurious falls in randomised controlled fall prevention trials: a systematic review. BMC Med Res Methodol. 2012 Apr 17;12:50. doi: 10.1186/1471-2288-12-50. PMID 22510239